CLINICAL TRIAL: NCT03771599
Title: The Effects of Traditional Massage on Spasticity and Activity of Children(2 to 10 Years) With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Qamar Mehmood, Senior Physiotherapist & Head of Physiotherapy Department NIRM, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIRS-IUISB/PHD/002
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Palsy, Spastic, Diplegic
Keywords: cerebral palsy, traditional massage, spasticity, children
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy; Muscle Spasticity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It is a RCT with two groups, control and intervention. Both groups received routine physical therapy five days a week for a period of three months. Intervention group also received traditional massage for thirty minutes before start of the routine physical therapy. Data was collected at baseline, after 06 weeks and 12 weeks of intervention
Who Masked: Outcomes Assessor
Masking Description: outcome assessor was kept blind about group identification of the participants before assessments at baseline, after 06 weeks and 12 weeks of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Routine physical therapy
  [Time Frame: Twelve weeks]
  Interventions: Other: Control group
- Intervention group (Experimental): Traditional massage + Routine physical therapy
  [Time Frame: Twelve weeks]
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Traditional massage of thirty minutes duration ( five minutes of massage was provided to all four limbs, front and back of trunk area) prior to routine physical therapy.
  Routine physical therapy comprising stretching of tight muscles ( stretch each muscle for five times with hold time of twenty seconds), Strengthening of weak muscles (perform resisted exercises ten times for each weak muscle), positioning ( how to make sitting and standing postures at home). This whole regimen was to be practiced fives times a week for a period of twelve weeks.
  Other Names: Routine physical therapy and Traditional massage
  Arms: Intervention group
Other: Control group — Routine physical therapy comprising stretching of tight muscles ( stretch each muscle for five times with hold time of twenty seconds), Strengthening of weak muscles (perform resisted exercises ten times for each weak muscle), positioning ( how to make sitting and standing postures at home). This whole regimen was to be practiced fives times a week for a period of twelve weeks.
  Other Names: Routine Physical Therapy
  Arms: Control group

SUMMARY:
The study has been conducted to see the effects of traditional massage on spasticity and activity of children with cerebral palsy (CP). It is a randomized controlled trial having two groups, control and intervention. Both groups received routine physical therapy treatment comprising stretching of tight muscles, strengthening of weak muscles, positioning and handling. Intervention group also received traditional massage in addition to routine physical therapy. Caregivers were trained to perform routine physical therapy treatment and traditional massage at home. Data was collected using a structured questionnaire, Modified Ashworth Scale (MAS), Gross Motor Function Classification System (GMFCS), Gross Motor Function Measure (GMFM) and CPChild Caregiver Priorities & Child Health Index of Life with Disabilities at baseline, after 06 weeks and 12 weeks of intervention.

DETAILED DESCRIPTION:
Physical therapy is an important component of rehabilitation regimen which is commonly used in the management of children with CP. Massage is also used as a complimentary alternative medicine (CAM). It has many types being practiced across the globe. Traditional massage is a type of massage being practiced in a specific society and has its own way of execution. It does not need professional education, training and certification so do not have any financial burden on the caregivers. As Pakistan is a poor country with low socio-economic status, so such measures of management which involve less financial burden on caregivers need to be investigated.

In this RCT, traditional massage was performed on the participants in the supine lying position. Each upper and lower limb was massaged for five minutes with gentle rubbing in proximal to distal direction. Five minutes massage was also provided at front and back of trunk area each in center to periphery direction. This type of traditional massage is practiced in Pakistan population which is somewhat different to Swedish massage. In few previous studies effect of Swedish massage on spastic CP has been investigated with conflicting level of evidence. However no study has been conducted in Pakistan to see the effects of traditional massage on children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Child should have diagnosis of spastic cerebral palsy (hemiplegic and diplegic types only).

Exclusion Criteria:

* Children having moderate to severe contractures.
* Children having moderate to severe mental retardation and with multiple disabilities.
* Children with Attention Deficit Hyperactive Disorder (ADHD), uncontrolled seizures and behavioral disorders

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth scale | Twelve weeks
  * 0 = No increase in muscle tone
  * 1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range Of Motion (ROM)
  * 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3 = Considerable increase in muscle tone, passive movement difficult.
  * 4 = Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
Gross motor Function Measure | Twelve weeks
  to see the gross motor ability having total of 88 items to be checked in 05 different domain Lying and Rolling (total score 51), Sitting (Total score 60), Crawling and Kneeling( total 42), standing (total 39), walking running jumping (total 72)
Gross Motor Function Classification System | Twelve weeks
  It has five levels I to V showing the mobility level. Level I to III represent ambulatory status while IV and V represent Non- ambulatory status
CPCHILD ( Caregiver Priorities & child health index of life with Disabilities | Twelve weeks
  to see the quality of life of children with cerebral palsy. It has 09 sections to be completed representing different states related to quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Isra University, Islamabad, Federal, Pakistan

REFERENCES:
- [Background] Reddihough DS, Collins KJ. The epidemiology and causes of cerebral palsy. Aust J Physiother. 2003;49(1):7-12. doi: 10.1016/s0004-9514(14)60183-5. PMID 12600249
- [Background] Kirby RS, Wingate MS, Van Naarden Braun K, Doernberg NS, Arneson CL, Benedict RE, Mulvihill B, Durkin MS, Fitzgerald RT, Maenner MJ, Patz JA, Yeargin-Allsopp M. Prevalence and functioning of children with cerebral palsy in four areas of the United States in 2006: a report from the Autism and Developmental Disabilities Monitoring Network. Res Dev Disabil. 2011 Mar-Apr;32(2):462-9. doi: 10.1016/j.ridd.2010.12.042. Epub 2011 Jan 26. PMID 21273041
- [Background] Bhasin TK, Brocksen S, Avchen RN, Van Naarden Braun K. Prevalence of four developmental disabilities among children aged 8 years--Metropolitan Atlanta Developmental Disabilities Surveillance Program, 1996 and 2000. MMWR Surveill Summ. 2006 Jan 27;55(1):1-9. PMID 16437058
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Paneth N, Hong T, Korzeniewski S. The descriptive epidemiology of cerebral palsy. Clin Perinatol. 2006 Jun;33(2):251-67. doi: 10.1016/j.clp.2006.03.011. PMID 16765723
- [Background] Reddihough DS, Jiang B, Lanigan A, Reid SM, Walstab JE, Davis E. Social outcomes of young adults with cerebral palsy. J Intellect Dev Disabil. 2013 Sep;38(3):215-22. doi: 10.3109/13668250.2013.788690. Epub 2013 May 14. PMID 23672634
- [Background] Goodman M, Rothberg AD, Houston-McMillan JE, Cooper PA, Cartwright JD, van der Velde MA. Effect of early neurodevelopmental therapy in normal and at-risk survivors of neonatal intensive care. Lancet. 1985 Dec 14;2(8468):1327-30. doi: 10.1016/s0140-6736(85)92626-1. PMID 2415788
- [Background] Hurvitz EA, Leonard C, Ayyangar R, Nelson VS. Complementary and alternative medicine use in families of children with cerebral palsy. Dev Med Child Neurol. 2003 Jun;45(6):364-70. doi: 10.1017/s0012162203000707. PMID 12785436
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350